CLINICAL TRIAL: NCT00823550
Title: A Randomized, Open Label, Phase IV, Multicenter Study for Efficacy and Safety of Lamivudine Versus Entecarvir Therapy in HBV-related Advanced Liver Disease Patients With High Viral Load and Normal or Slightly Elevated Transaminase
Brief Title: Antiviral Therapy in Hepatitis B Virus (HBV)-Related Advanced Liver Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Kangbuk Samsung Hospital (Other); Konkuk University Hospital (Other); Chung-Ang University (Other); Ajou University (Other); Inha University Hospital (Other); Soonchunhyang University Hospital (Other); The Catholic University of Korea (Other); Hallym University Medical Center (Other); Kyungpook National University Hospital (Other); Keimyung University (Other); Korea University Anam Hospital (Other); Korea University (Other); Hanyang University (Other); Inje University (Other); Pusan National University Hospital (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Kwang-Hyub Han, Department of Internal Medicine, Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0296
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2009-01

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; Advanced fibrosis; Lamivudine; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): entecavir 0.5 mg QD
  Interventions: Drug: Entecavir
- B (Active Comparator): lamivudine 100 mg QD
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — entecavir 0.5 mg QD
  Other Names: Baraclude 0.5mg
  Arms: A
Drug: Lamivudine — lamivudine 100 mg QD
  Other Names: Zeffix 100mg
  Arms: B

SUMMARY:
This is a randomized, open label, phase IV, multicenter study for efficacy and safety of lamivudine versus entecarvir therapy in HBV-related advanced liver disease patients with high viral load and normal or slightly elevated transaminase.

DETAILED DESCRIPTION:
Currently, treatment guidelines for the management of chronic hepatitis B (CHB) recommend that patients with serum HBV DNA > 105 copies/ml and elevated ALT levels greater than two times the upper limit of normal (ULN) are obvious candidates for antiviral therapy. Guidelines also suggest that antiviral therapy be considered in CHB patients with high viral load, if a biopsy shows significant liver disease despite ALT ≤ 2× ULN. Data from recent trials in hepatitis B patients who present with normal to minimally elevated ALT (≤ 2× ULN) indicate that significant hepatic pathology could still be found. Serum ALT level may not accurately predict activity of liver damage. ALT is a poor predictor of outcome and therefore is not a suitable criterion for antiviral therapy in chronic hepatitis B infection. Also, a recent large randomized controlled clinical trial comparing lamivudine maintenance and placebo in advanced fibrosis (Ishak fibrosis score ≥ 4) suggests that sustained viral suppression with antiviral therapy is linked to reduced risk for disease progression. (Liaw YF et al. NEJM 2004;351:1521-1531)

ELIGIBILITY:
Inclusion criteria

* Male and female, 18 years of age or older
* HBsAg positive for more than 6 months
* Serum HBV DNA > 2,000 IU/ml
* Serum ALT < 2 X ULN on two consecutive occasions at least 3 months apart
* Naïve to nucleoside or nucleotide therapy
* On liver biopsy, fibrosis score ≥ 3 according to METAVIR scoring system (within 2 years of Day 0)
* If liver biopsy is not available, subjects must have two of the following items

  * Overt findings of cirrhosis by radiologic evidence (MRI, CT, US)
  * Gastrointestinal varices
  * Platelet count < 100,000,Splenomegaly (Spleen size - 12cm)
* The patient who is willing and able to provide written informed consent to participate in this study

Exclusion criteria

* A history of SBP, variceal bleeding, HEP, HCC
* Decompensated liver disease (Child-Pugh score > 10)
* Co-infected with HCV or HIV
* History of any other forms of liver disease.
* Patient who is pregnant or breastfeeding
* Treatment with immunosuppressive, immunomodulatory agents or antiviral agents within 6 months prior to study entry
* A history of liver transplantation or planned for liver transplantation
* A history of any other medical disease or condition that would make the patients unsuitable for the study.
* Patient is currently abusing alcohol or illicit drugs or has a history of alcohol abuse or illicit substance abuse within the preceding 2 years.
* Patient is enrolled or plans to enroll in another clinical trial of an investigational agent while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression as defined by the first occurrence of any of the cirrhosis compolications | 5 years

SECONDARY OUTCOMES:
Proportion of patients achieving either HBV DNA level ≤ 60 IU/mL Proportion of patients with ALT normalization Proportion of patients with HBeAg loss and seronconversion Proportion of patients with virologic breakthrough | at months 12, 24, 36, 48, and 60

CONTACTS AND LOCATIONS:
Overall Officials: Kwnag-Hyub Han, MD, Study Chair — Yonsei Univsersity College of Medicine; Jun Yong Park, MD, Study Director — Yonsei Univsersity College of Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea